CLINICAL TRIAL: NCT04801511
Title: Safety and Efficacy of Preoperative IMRT (Intensity-modulated Radiation Therapy) With Concurrent High-dose Intravenous Vitamin C and mFOLFOX6 in Locally Advanced Rectal Cancer Patients: a Prospective Study.
Brief Title: Preoperative IMRT With Concurrent High-dose Vitamin C and mFOLFOX6 in Locally Advanced Rectal Cancer
Acronym: CORT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhou Fuxiang (Other)
Responsible Party: Sponsor-Investigator, Zhou Fuxiang, professor, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCCSC R02
Record Dates: First submitted 2021-03-11; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; neoadjuvant; chemoradiotherapy; Vitamin C
MeSH Terms: conditions — Rectal Neoplasms | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Preoperative CRT: The eligible subjects will be treated with concurrent chemoradiotherapy and high-dose intravenous vitamin C. IMRT will be delivered to PTV-CTV (plan target volume-clinical target volume) with a dose of 45Gy/25f. If necessary, additional boost of 5-10Gy will be delivered to PTV-GTV (plan target volume- gross tumor volume). During the IMRT, 2-3 cycles of concurrent chemotherapy (mFOLFOX6) will be delivered. High-dose intravenous vitamin C (24g/d，QD) will be delivered on the day of radiotherapy from the beginning to the end. Three additional cycles of chemotherapy (mFOLFOX6) will be given after radiotherapy. Radical surgery will be performed approximately 10-12 weeks after the end of radiotherapy. Whether or not to select "watch and wait" or sphincter preserving surgery needs to refer to the tumor location, tumor regression, surgeon's opinion and patient's will.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Preoperative concurrent chemoradiotherapy and high-dose intravenous vitamin C :
  The eligible subjects will be treated with concurrent chemoradiotherapy and high-dose intravenous vitamin C preoperatively. IMRT will be delivered to PTV-CTV (plan target volume-clinical target volume) with a dose of 45Gy/25fraction/5weeks. If necessary. During IMRT, 2-3 cycles of concurrent chemotherapy (mFOLFOX6) will be delivered. High-dose intravenous vitamin C ( 24g/d，QD ) will be delivered on the day of radiotherapy from the beginning to the end of IMRT.
  preoperative consolidation chemotherapy: Three additional cycles of neoadjuvant chemotherapy (mFOLFOX6) will be given after the end of IMRT.
  TME （total mesorectal excision）or sphincter preserving surgery will be performed approximately the 10th-12th weeks after the end of IMRT. Whether or not to select "watch and wait" needs to refer to the tumor location, tumor regression, surgeon's opinion and patient's will.
  Interventions: Drug: Vitamin C

INTERVENTIONS:
Drug: Vitamin C — High-dose Intravenous Vitamin C will be delivered on the day of radiotherapy, in order to reduce the acute toxicity of chemoradiotherapy.
  Other Names: ascorbic acid

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of preoperative chemoradiotherapy (IMRT) with concurrent high-dose intravenous vitamin C and mFOLFOX6 in locally advanced rectal cancer patients.

DETAILED DESCRIPTION:
Sixty patients with locally advanced rectal cancer (cT3-4N0M0, cT1-4N1-2M0, ≤12cm from anus) will be enrolled and receive preoperative IMRT concurrent with high-dose intravenous vitamin C and 2-3 cycles of mFOLFOX6 chemotherapy, and then after 4 weeks rest, they will continue to complete 3 cycles of preoperative chemotherapy (mFOLFOX6). Radical surgery will be performed at 10-12 weeks after IMRT.

In this study, we will evaluate the safety and effectiveness of the treatment method through the acute toxicity [during CRT (concurrent chemoradiotherapy )], PCR (pathologic complete response) rate, sphincter preserving surgery rate, 2-year survival rate and 2-year disease-free survival rate.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years of age with a confirmed histopathologic diagnosis of adenocarcinoma of the rectum and considered suitable for curative resection.
2. Tumors were clinically confirmed (by MRI or CT plus endorectal ultrasound) as stage II (cT3-4N0) or stage III (cT1-4N1-2), with a positive node defined as ≥1.0 cm in diameter on imaging) and a distal border located , 12 cm from the anal verge.
3. Patients were required to have an Eastern Cooperative Oncology Group performance status ≤ 1 and adequate hematologic, liver, and renal function. (HGB≥90g/L, WBC≥3.5×10^9/L, PLT≥90×10^9/L；ALT / AST≤2.5× ULN；T BILL≤1.5×ULN，Cr ≤1.5×ULN)
4. Laboratory examination showed that glucose-6-phosphate dehydrogenase (G6PD) was normal.
5. The patient agreed and had signed the informed consent

Exclusion Criteria:

1. With metastatic disease.
2. Prior radiotherapy or chemotherapy.
3. The presence of other cancers.
4. Clinically significant cardiac disease.
5. Known peripheral neuropathy.
6. With intestinal obstruction, intestinal perforation or tumor bleeding who need emergency operation.
7. Rectal cancer with signet-ring cell carcinoma, or with Neuroendocrine tumor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-08 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PCR rate | 2 year From the first subject underwent surgery to the last subject underwent surgery.
  The PCR rate is defined as the percentage of subjects who achieved Pathological complete remission（PCR） in the total number of the subjects who underwent surgery in the ITT population.

SECONDARY OUTCOMES:
acute toxicity | 2 year
  acute toxicity including diarrhea， vomiting leukopenia, er al, during the preoperative CRT and high-dose intravenous vitamin C and 30 after the radiotherapy.
Resection rate of anus preserving surgery | 2 year From the first subject underwent surgery to the last subject underwent surgery.
  In patients with low rectal cancer, the percentage of subjects who underwent anus preserving surgery accounted for the total TME surgery.
2-year survival rate | up to 2 years after the last subject being enrolled
  2-year survival rate of ITT (Intent to treat) population.
2-year disease-free survival rate | up to 2 years after the last subject being enrolled.
  2-year disease-free survival rate of ITT population.

CONTACTS AND LOCATIONS:
Overall Officials: Fuxiang Zhou, M.D., Study Chair — Zhongnan Hospital
Locations (1):
- Zhongnan Hopital of Wuhan University, Wuhan, Hubei, China